CLINICAL TRIAL: NCT01900756
Title: Tailored Hospital-based Risk Reduction to Impede Vascular Events After Stroke
Acronym: THRIVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1U01NS079179 (NIH)
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral (Active Comparator): 1. Pre-appointment phone text
  2. In-clinic educational video
  3. Patient report card
  4. Post-clinic phone text
  5. Outpatient stroke registry
  Interventions: Behavioral: THRIVES
- Standard care (No Intervention): Routine and customary management.

INTERVENTIONS:
Behavioral: THRIVES — Pre-appointment phone text In-clinic educational video Patient report card Post-clinic phone text Outpatient stroke registry
  Arms: Behavioral

SUMMARY:
The purpose of this study is to determine whether a culturally-sensitive multipronged post-discharge intervention can significantly reduce blood pressure, enhance achievement of guideline recommended targets for risk factor control, and lower recurrent vascular events in a low-income and middle-income (LMIC). The study will have 2 Phases - a qualitative phase (Phase 1) lasting less than one year involving development of the intervention through focus group methodologies and structured interviews, and a clinical trial phase (Phase 2)lasting 3 years involving a randomized trial testing the efficacy of the intervention.

DETAILED DESCRIPTION:
This research seeks to develop an effective and sustainable way of reducing the devastating and deadly impact of stroke in a low-income region of the world with poor medical infrastructure. It will do so by focusing on improving the treatment of the condition most closely tied to stroke, hypertension, using novel methods that incorporate the input of the local community. If successful, the strategy could serve as a ready model to be adapted by decision-makers in other under-resourced areas for lessening the burden of stroke(and other major public health challenges).

ELIGIBILITY:
Phase 1: Inclusion Criteria:

Age ≥ 18 years Stroke within one year access to mobile phone.

Exclusion Criteria:

Any medical condition that would limit participation in follow up assessments, Severe cognitive impairment/dementia (MMSE ≤24) Severe global disability (modified Rankin Score ≥ 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Reduction in systolic blood pressure | 1 year
  Reduction in systolic blood pressure at one year post-discharge in stroke patients.

SECONDARY OUTCOMES:
Reduced rate of subsequent primary vascular event | 1 year

OTHER OUTCOMES:
Reduction of disability and enhanced quality of life. | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- Nigeria (3):
  - Sacred Heart Hospital, Abeokuta, Ogun State
  - Federal Medical Centre, Abeokuta
  - University College Hospital, Ibadan

REFERENCES:
- [Derived] Owolabi MO, Gebregziabher M, Akinyemi RO, Akinyemi JO, Akpa O, Olaniyan O, Salako BL, Arulogun O, Tagge R, Uvere E, Fakunle A, Ovbiagele B. Randomized Trial of an Intervention to Improve Blood Pressure Control in Stroke Survivors. Circ Cardiovasc Qual Outcomes. 2019 Dec;12(12):e005904. doi: 10.1161/CIRCOUTCOMES.119.005904. Epub 2019 Dec 6. PMID 31805787
- [Derived] Owolabi MO, Akinyemi RO, Gebregziabher M, Olaniyan O, Salako BL, Arulogun O, Ovbiagele B. Randomized controlled trial of a multipronged intervention to improve blood pressure control among stroke survivors in Nigeria. Int J Stroke. 2014 Dec;9(8):1109-16. doi: 10.1111/ijs.12331. Epub 2014 Jul 18. PMID 25042605